CLINICAL TRIAL: NCT06337890
Title: The Use of CO2 Automated Angiographies Combined With Fusion Imaging to Obtain Zero- or Near Zero- Contrast FEVAR for Complex Aortic Aneurysms.
Brief Title: CO2 Automated Angiographies With Fusion Imaging for Zero- or Near Zero- Contrast FEVAR.
Status: Recruiting | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Enrico Gallitto, Principal Investigator, University of Bologna
Other Study IDs: FEZECO
Record Dates: First submitted 2024-03-18; First posted 2024-03-29 (Actual); Last update posted 2024-03-29 (Actual); Status verified 2024-03

CONDITIONS: Aortic Aneurysm
Keywords: FEVAR; CO2; Complex aortic aneurysm
MeSH Terms: conditions — Aortic Aneurysm

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CO2 FEVAR: Use of automated CO2 angiographies combined with Fusion Imaging in patients with complex aortic aneurysms to obtain zero- or near zero- contrast FEVAR
  Interventions: Procedure: Zero contrast FEVAR

INTERVENTIONS:
Procedure: Zero contrast FEVAR — Use of automated CO2 angiographies with Fusion Imaging for zero contrast FEVAR

SUMMARY:
Fenestrated endovascular aneurysm repair (FEVAR) is an established technique used to treat complex aortic aneurysms (TAAAs), with satisfactory early and midterm results.

Postoperative renal function worsening is a common adverse event after FEVAR of complex aneurysms and is associated with prolonged hospital stay, higher morbidity, and long-term mortality in the peri-operative period and during follow-up. One of the more common causes of renal function worsening is contrast-induced nephropathy resulting from the use of iodinated contrast medium (ICM).

Automated carbon dioxide (CO2) angiography has been proposed as an alternative to ICM for standard endovascular aneurysm repair (EVAR) in consideration of its absence of nephrotoxicity that can be of further help in preserving renal function.

In adjunct, hybrid room and fusion imaging (FI) technologies are useful tools to reduce intraoperative contrast medium and fluoroscopy time.

In literature there are few reports regarding the use of CO2 for fenestrated endografting repair of complex aortic aneurysms.

The aim of the present study is to report the possibility to combine the use of automated CO2 angiographies and Fusion Imaging to obtain zero- or near zero- contrast FEVAR for complex aortic aneurysms.

DETAILED DESCRIPTION:
Fenestrated endovascular aneurysm repair (FEVAR) is an established technique used to treat juxtarenal and pararenal abdominal aortic aneurysms (AAAs) and type IV thoracoabdominal aortic aneurysms (TAAAs), as demonstrated by early and midterm literature results.

Postoperative renal function worsening is a common adverse event after FEVAR of complex aneurysms and is associated with prolonged hospital stay, higher morbidity, and long-term mortality in the peri-operative period and during follow-up.

Renal function may worsen after FEVAR because of a variety of factors, but one of the more common causes of renal function worsening is contrast-induced nephropathy resulting from the use of iodinated contrast medium (ICM).

Automated CO2 angiography has been proposed as an alternative to ICM for standard endovascular aneurysm repair (EVAR) in consideration of its absence of nephrotoxicity that can be of further help in preserving renal function.

In adjunct, hybrid room and fusion imaging (FI) technologies, based on a three-dimensional preoperative computed tomography angiography (CTA) image over-laid on a two-dimensional live fluoroscopy image, are useful tools to reduce intraoperative contrast medium and fluoroscopy time.

The aim of the present study is to report the possibility to combine the use of automated CO2 angiographies and Fusion Imaging to obtain zero- or near zero- contrast FEVAR for complex aortic aneurysms.

ENDPOINTS

Early: - Technical success (defined as correct endograft deployment with stenting and patency of all planned target visceral vessels (TVVs) and absence of type I and type III endoleaks, iliac leg stenosis or kinking and mortality at 24 hours)

* in-hospital/30-day reintervention and mortality
* perioperative renal function worsening (according to the RIFLE, Risk, Injury, Failure, Loss of kidney function, End-stage renal disease, criteria)

Follow-up: - Freedom from TVVs instability

* Survival
* Freedom from reintervention
* Freedom from renal function worsening

CO2 Injection protocol

Diagnostic CO2 angiographies are performed in the anteroposterior and 90-degree lateral projections from a 6F sheet, positioned in the pararenal aorta, by an automated CO2 injector (Angiodroid; San Lazzaro, Bologna, Italy).

The FI/VesselNavigator is optimized with these two CO2 angiography images and the TVV origins. The injection pressure and volume are usually set at 650 mmHg and 100 ml, respectively. Carbon dioxide angiographies are repeated step by step after endograft introduction and during endograft deployment to adjust the endograft's position according to fusion images.

To evaluate cannulation and bridging stentgraft deployment in each TVVs CO2 angiographies are performed with the 6F sheet for superior mesenteric artery and, for the other TVVs, with selective angiographies through the TVVs sheet.

In this case, the injection pressure is set at 300 mmHg while the injection volume is set at 40 mL.

The angiographic shots required to deploy the bifurcated graft and the contralateral iliac leg are usually performed through an automated CO2 injection from the femoral sheaths.

Completion angiography is performed through 6F sheet positioned in the proximal portion of the endograft, in both anteroposterior and lateral views.

FOLLOW-UP

30-day: CTA scan + blood tests 3 months: duplex ultrasound (DUS) or CTA scan (in case of any doubt) + blood tests 6 months: DUS + blood tests 12 months: CTA scan + blood tests

During the follow-up, clinical evaluations will be performed as per standard clinical practice for patients with this condition.

ELIGIBILITY:
Inclusion Criteria:

* Patients with complex aortic aneurysms eligible for FEVAR.
* Obtaining informed consent.
* Age >18 years at the time of diagnosis

Exclusion Criteria:

* Age <18 years at the time of diagnosis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All the patients with complex aortic aneurysms (according to SVS guidelines) that undergo FEVAR with automated CO2 angiographies combined with Fusion Imaging to reduce the amount of iodinated contrast medium
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of technical success | 24-hour
  correct endograft deployment with stenting and patency of all planned TVVs and absence of type I and type III endoleaks, iliac leg stenosis or kinking and mortality at 24 hours
Reintervention and mortality | 30-day
  In-hospital/30-day
Number of participants with perioperative renal function worsening | 30-day
  according to RIFLE classification
Rate of TVVs instability | through study completion, an average of 1 year
  Freedom from TVVs instability
Rate of survival | through study completion, an average of 1 year
  Survival
Rate of reintervention | through study completion, an average of 1 year
  Freedom from reintervention
Number of participants with renal function worsening | through study completion, an average of 1 year
  Freedom from renal function worsening

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Gallitto, Principal Investigator — University of Bologna
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy